CLINICAL TRIAL: NCT06243159
Title: JY231 Injection for the Treatment of Refractory Autoimmune Diseases (ADs) Early Exploratory Clinical Studies on Safety, Tolerability, and Initial Efficacy
Brief Title: JY231(Internal Clinical Drug Code) Injection for the Treatment of Refractory Autoimmune Diseases
Acronym: JY231、ADs
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanxi Bethune Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JY-CT-23-007
Record Dates: First submitted 2024-01-26; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Autoimmune Diseases
Keywords: JY231 injection
MeSH Terms: conditions — Autoimmune Diseases | interventions — fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JY231 injection for the treatment of refractory autoimmune diseases (ADs) Early exploratory clinica (Experimental): Infusion of JY231 Injection by dose of 1-10×10^6 transducing units(TU)/kg、 1-5×10^7 TU/kg、5-10 ×10^7 TU/kg Administration method: intravenous infusion、Splenic artery infusion、Lymph node infusion; Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion (PI evaluation is required)
  Interventions: Genetic: JY231

INTERVENTIONS:
Genetic: JY231 — Infusion of JY231 Injection by dose of 1-10×10^6 TU/kg、 1-5×10^7 TU/kg、5-10 ×10^7 TU/kg Administration method: intravenous infusion、Splenic artery infusion、Lymph node infusion; Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion (PI evaluation is required)
  Other Names: Fludarabine; Cyclophosphamide

SUMMARY:
Early exploratory clinical study of the safety, tolerability and initial efficacy of JY231 injection in the treatment of refractory autoimmune diseases

DETAILED DESCRIPTION:
This is a single-center, single-arm. open-treatment clinical study, in this study. approximately 10-20 adult and elderly patients with refractory autoimmune diseases will be enrolled for JY231 infusion therapy. The safety of JY231 was evaluated by observing adverse events after cell therapy. Evaluate the effectiveness of JY231 treatment compared to the results of the subjects' own previous standard treatment regimens or base data.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65 years old, regardless of gender, signed with informed consent (ICF).
2. Diagnosed as one of the following diseases: Systemic lupus erythematosus (SLE)；Sjogren's syndrome (SS) ; Systemic Scleroderma (SSc); Dermatomyositis (DM); Anti neutrophil cytoplasmic antibody associated vasculitis (ANCA-AAV).
3. Patients who have been treated with ≥ 2 immunosuppressive agents for 3 months, or require ≥ 15mg glucocorticoids to maintain stable condition, or are intolerant to standard treatment, or have relative contraindications, and whose disease activity meets the following criteria:

   1. For SLE patients, SLEDAI ≥ 8 points;
   2. For SS patients, Sjogren's syndrome disease activity index(ESSDAI )≥ 14 points;
   3. For SSc patients, the modified Rodnan skin score (mRSS) score ranges from 10 to 35 (including cutoff values) and is associated with interstitial pneumonia (ILD);
   4. For DM patients, diagnosed for at least 1 year;
   5. For ANCA-AAV patients, Birmingham Vasculitis Activity Score(BVAS) score ≥ 15 and ANCA antibodies.
4. Eastern Cooperative Oncology Group(ECOG) 0-1 points;
5. The evaluation of important organ functions meets the following conditions:

   1. Blood count: hemoglobin ≥ 60g/L, platelet count ≥ 30 × 109/L;
   2. Cardiac function: Left ventricular ejection fraction (LVEF) ≥ 55%, no significant abnormalities observed on electrocardiogram;
   3. Renal function: estimated glomerular filtration rate(eGFR) ≥ 30 mL/min/1.73m2;
   4. Liver function: Aspartate Aminotransferase(AST) and Alanine Transaminase(ALT) ≤ 3.0 upper limit of normal(ULN), total bilirubin ≤ 2.0 ULN;
   5. Pulmonary function: diffusion capacity of the lung for carbon monoxide(DLCO) ≥ 40% expected value; forced vital capacity(FVC) ≥ 50% of expected value;
   6. Having single or intravenous blood collection standards and no other contraindications for cell collection;
6. The urine pregnancy test results of subjects of childbearing age are negative, and they agree to take effective contraceptive measures during the trial period, until one year after infusion;
7. The patient or their guardian agrees to participate in this clinical trial and signs an informed consent form, indicating their understanding of the purpose and procedures of this clinical trial and willingness to participate in the study.

Exclusion Criteria:

1. Previously received Chimeric Antigen Receptor T cell(CAR-T) therapy;
2. Suffering from severe diseases of the heart, liver, lungs, blood system, and endocrine system, the researcher has determined that the risk of participating in the trial is higher than the benefit;
3. Active or uncontrollable infections that require systemic treatment within the first week of screening;
4. Previously received hematopoietic stem cell transplantation or solid organ transplantation (excluding corneal and hair transplantation), or screened for acute graft-versus-host disease (GVHD) with grade 2 or above in the first two weeks;
5. Hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) is positive and the hepatitis B virus(HBV) DNA titer in peripheral blood is greater than the normal reference value; Or hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA titer detection greater than the normal reference range; Or positive for human immunodeficiency virus (HIV) antibodies; Or those who test positive for syphilis; Or positive for cytomegalovirus (CMV) DNA detection;
6. Received live vaccine within 4 weeks prior to screening;
7. Pregnancy test positive individuals;
8. Patients with malignant tumors and other malignant diseases before screening, in addition to fully treated cervical cancer in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical surgery, and ductal carcinoma in situ after radical surgery;
9. Screening patients who have participated in other clinical trials within the first three months;
10. Other researchers believe that it is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-08 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Day 0、Month 1、Month 2、Month 3、Month 6、Month 12
  Metric/method of measurement: (2007)《Revised response criteria for malignant lymphoma》

CONTACTS AND LOCATIONS:
Overall Officials: liyun zhang, Doctoral, Principal Investigator — Shanxi Bethune Hospital
Locations (1):
- Shanxi Bethune Hospital, Taiyuan, Shanxi, China